CLINICAL TRIAL: NCT03969342
Title: Standardization of Mid-Level Providers Using Point of Care Ultrasound to Diagnose Pediatric Pneumonia
Acronym: POCUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bridge to Health Medical and Dental (Other)
Collaborators: University of Toronto (Other); Kigezi Healthcare Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2
Record Dates: First submitted 2019-05-10; First posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Pneumonia; Pediatric Disorder; Diagnostic and Monitoring Radiological Devices Associated With Adverse Incidents
Keywords: Pediatric; Pneumonia; Ultrasound; Point of Care Ultrasound; Diagnostic Imaging; Global Health; Uganda; Rural Healthcare
MeSH Terms: conditions — Pneumonia; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Trainees (Experimental): Local mid-level providers who undergo five day training on point of care ultrasound for diagnosing pediatric pneumonia
  Interventions: Device: Point of care ultrasound training

INTERVENTIONS:
Device: Point of care ultrasound training — Five-day in-person training on point of care ultrasound using portable ultrasound devices followed by remote monitoring of practice scanning

SUMMARY:
The POCUS training program aims to bring sustainable, affordable access to POCUS to patients in need of diagnostic services in Uganda. This research study seeks to demonstrate that Clinical Officers (COs) in rural Uganda can be trained on POCUS for pediatric pneumonia, and that this training can be completed through remote monitoring and observation.

DETAILED DESCRIPTION:
Objectives To prove that mid-level providers in low-resource settings can be trained to use POCUS to diagnose pediatric pneumonia through a five-day training program followed by six months of remote analysis.

Study Design and Methods The investigators propose a remote evaluation study assessing the ability of POCUS program trainees in Kabale to obtain and evaluate pediatric lung scans. The indicator of interest will be diagnosis of pneumonia or lack thereof.

Trainee Selection:

Trainees were selected from the pool of mid-level providers who work with Kigezi Healthcare Foundation (KIHEFO) and who participated in needs assessment questionnaires in February 2018. From those respondents who indicated that they would like to participate in the training program, seven were selected based on their work ethic and their likelihood of working in the Kabale region for the foreseeable future.

Data Collection, Management, and Sharing:

Scanning will take place during the KIHEFO clinics in town and outreach. As well, some scanning may take place during the Bridge to Health Medical and Dental (BTH) and KIHEFO partnered brigade. Additionally, some scans will be collected at the Kabale Regional Referral Hospital.

KIHEFO is a Ugandan registered non-profit organization and a rural teaching site of Mbarara University of Science and Technology. KIHEFO has organized all brigades for the past six years and regularly conducts outreach clinics through a grant provided by the Ugandan Government and USAID.

Trainees will ask to conduct an ultrasound scan for practice on pediatric (under 18 years) patients with a cough, fever, and/or increased work of breathing. To avoid the possibility of trainees diagnosing patients based on scans, trainees will not scan their own patients, but rather, the patients of their peers. Ultimately, all trainees are Ugandan clinicians and licensed and regulated by appropriate Ugandan agencies. While the investigators cannot confirm that clinicians will act with integrity at all times, the investigators rely on the good training and integrity of the trainees as well as the relevant Ugandan health agencies to monitor care of patients.

Should the patient provide informed consent, while scanning, the trainee will fill out a case report form (CRF). The patient will be assigned an anonymous patient identification (ID) number, and trainees have each received a unique trainee ID number in order to conceal their identity from reviewers and maintain a blind study.

Scans and CRFs will be uploaded to an online "cloud." Each time a reviewer accesses a scan from the cloud, the reviewer will fill out a CRF. The CRFs of the trainee and the reviewer will later be compared to determine agreement or disagreement. As well, the trainee will record their clinical management and whether or not antibiotics were prescribed. This clinical information will be managed by the study coordinator.

Once trainees reach a predetermined level of agreement with expert reviewers, trainees will be considered standardized and permitted to use POCUS to diagnose pneumonia.

Ethical Consideration:

Expert reviewers will be blinded as to the identity of the trainees while reviewing scans; this will ensure that reviewers remain impartial while reading images.

Patient identifying information will not be disclosed to reviewers, or to any other non-essential parties. Each patient will be assigned an ID number upon receiving a scan, which is used when uploading the scan and on the CRF. Should a reviewer have a concern about a patient, the reviewer can give the patient's ID number to the local coordinator in Uganda, who has a coded list of patient information. The local coordinator can use this information to get in touch with the patient.

Until they are standardized, trainees are not experts in POCUS, and are not allowed to use POCUS to diagnose patients. All patients will receive a standard examination, and will be diagnosed and treated as usual before being asked to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Mid-level provider working in Kabale, Uganda
* Participated in pre-program needs assessment
* Able to continue practicing POCUS in Kabale through the duration of the study

Exclusion Criteria:

* Inability to continue practicing POCUS in Kabale through the duration of the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Trainee Scan Acquisition | 7 months
  The frequency at which trainees are able to acquire high-quality pediatric lung scans.
Trainee / Reviewer Diagnostic Agreement | 9 months
  The extent to which agreement between the diagnoses provided by our trainees, and that provided by our expert reviewers, is statistically significant.

CONTACTS AND LOCATIONS:
Overall Officials: William Cherniak, BSc, MD, MPH, CCFP(EM), DABFM, Principal Investigator — Bridge to Health Medical and Dental
Locations (1):
- Kigezi Healthcare Foundation (KIHEFO), Kabale, Uganda

IPD SHARING:
Plan to Share IPD: No
No Individual Participant Data (IDP) sharing plan.